CLINICAL TRIAL: NCT01892254
Title: Inkretineffekten Hos Patienter Med Polycystisk Ovariesyndrom før og Efter Behandling af Insulinresistens (Incretin Effect in Patients With Polycystic Ovary Syndrome Before and After Treatment of Insulin Resistance)
Brief Title: Incretin Effect in PCOS Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Louise Vedtofte, Humanbiolog, ph.d., University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PCOS-INK
Record Dates: First submitted 2013-06-11; First posted 2013-07-04 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: incretin effect; PCOS; insulin resistance; OGTT; IIGI
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin-Placebo (Experimental): Metformin, 2x 2 tablets a day, 500 mg tablets for 12 weeks, 6 weeks wash-out, 12 weeks placebo
  Interventions: Drug: Metformin; Drug: Placebo
- Placebo-metformin (Placebo Comparator): Placebo tablets, 2x 2 tablets per day for 12 weeks, 6 weeks wash-out, 12 weeks metformin, 2x 2 tablets per day, 500 mg per tablet
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin, 2x 2 tablets a day, 500 mg tablets
  Other Names: 657-24-9
Drug: Placebo — Placebo (to metformin)

SUMMARY:
This study investigates the incretin effect in women with polycystic ovary syndrome (PCOS) before and after removal of their insulin resistance by metformin.

The investigators' hypothesis is that insulin resistant women with PCOS have a reduced incretin effect and elevated glucagon responses as measured by a 75-g oral glucose tolerance test and isoglycemic i.v. glucose infusion. The investigators hypothesise that both can be improved when their insulin resistance is removed.

ELIGIBILITY:
Inclusion Criteria PCOS-women:

* Diagnosed with PCOS according to the Rotterdam criteria
* more than 18 years old
* BMI less than 30 kg/m2
* Normal glucose tolerance and fasting plasma glucose (assessed by 75-g OGTT)
* Negative GAD65 and islet cell autoantibodies
* Insulin resistant according to HOMA-IR
* informed consent

Inclusion Criteria healthy women:

* more than 18 years old
* BMI less than 30 kg/m2
* Normal glucose tolerance and fasting plasma glucose (assessed by 75-g OGTT)
* Negative GAD65 and islet cell autoantibodies
* informed consent
* regular menstrual cycle (28-35 days)
* Plasma androgen levels within reference levels

Exclusion Criteria PCOS and healthy women:

* First or second degree relatives with diabetes
* pregnancy or breast feeding
* treatment with medication which influences the glucose metabolism (incl hormonal contraception)
* Congenital diseases which cause hyperandrogenism and irregular bleeding
* Known adrenal hyperplasia
* Known hyperprolaktinemia
* Alcohol consumption of more than 20 grams a day
* Hemoglobin less than 7.8 %

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
The change in incretin effect from baseline and until after removal of insulin resistance | baseline and 12 weeks' treatment
  The incretin effect will be assessed from the insulin secretion during af 75 g OGTT and IIGI at baseline and after 12 weeks' treatment with placebo and metformin

SECONDARY OUTCOMES:
Glucagon response | 0, 12 and 30 weeks
  Glucagon responses (plasma concentrations) will be assessed during the 75-g OGTTs

CONTACTS AND LOCATIONS:
Overall Officials: Louise Vedtofte, MSc., PhD, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (1):
- Copenhagen University Hospital Gentofte, Hellerup, Select A State, Denmark